CLINICAL TRIAL: NCT03419663
Title: Cereal or Grain Consumption and Gastric Cancer Risk: a Systematic Review and Meta-analysis of Observational Studies
Brief Title: Systematic Review and Meta-analysis of Cereal or Grain Consumption and Gastric Cancer
Acronym: GC
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong Zhou, associate chief physician, West China Hospital
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Gastric Cancer
Keywords: cereal; whole grain; refined grain; gastric cancer; meta analysis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Edible Grain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- gastric cancer
  Interventions: Dietary Supplement: cereal or grain consumption

INTERVENTIONS:
Dietary Supplement: cereal or grain consumption — intake of cereal, whole grain, refined grain, and other grain of every day

SUMMARY:
This project involved a systematic literature review of published trials of cereal or grain in relation to the risk of gastric cancer. Data was extracted from the publications on PubMed, EMBASE, Cochrane Library.A traditional meta-analysis, subgroup analysis, and heterogeneity was conducted on the extracted data.

DETAILED DESCRIPTION:
Investigators searched PubMed, EMBASE, Cochrane Library for studies focusing on cereal or grain in relation to the risk of gastric cancer up to October 2017. Summary odd ratios (OR) and 95% confidence intervals (CI) were calculated by using either random effect models or fixed effect models according to the heterogeneity of included studies. Subgroup analysis, heterogeneity, and publication bias were also performed.

ELIGIBILITY:
Inclusion Criteria:

* a case-control studies or a cohort study
* investigate the association between cereal or grain intake and GC occurrence
* report an odds ratio (OR) or relative risk (RR) with corresponding 95% confidence intervals (CI)
* provide sufficient data to estimate OR or RR

Exclusion Criteria:

* Non-human studies
* GC mortality-based cohort studies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, both children and adults, regardless of health status
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
the relationship between overall cereal consumption and gastric cancer occurance | up to 2 years
  perform a pooled analysis of included studies with OR through STATA 12.0

SECONDARY OUTCOMES:
the relationship between whole grain and gastric cancer occurance | up to 2 years
  perform a subgroup analysis to summarize the related OR through STATA 12.0
the relationship between refined grain and gastric cancer occurance | up to 2 years
  perform a subgroup analysis to summarize the related OR through STATA 12.0
the relationship between other grain and gastric cancer occurance | up to 2 years
  perform a subgroup analysis to summarize the related OR through STATA 12.0

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Xu Y, Yang J, Du L, Li K, Zhou Y. Association of whole grain, refined grain, and cereal consumption with gastric cancer risk: A meta-analysis of observational studies. Food Sci Nutr. 2018 Nov 11;7(1):256-265. doi: 10.1002/fsn3.878. eCollection 2019 Jan. PMID 30680179

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03419663/SAP_001.pdf